CLINICAL TRIAL: NCT07152327
Title: Effectiveness of Terbinafine Hydrochloride in the Treatment of Otomycosis: Basic and Clinical Evaluation
Brief Title: Terbinafine Hydrochloride for the Treatment of Otomycosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Samy Mohamed Abd Ellatief, resident , ENT, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTO-Terbinafine-2025
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Otomycosis; Fungal Ear Infection
Keywords: Otomycosis; Aspergillus; Candida
MeSH Terms: conditions — Otomycosis; Torulopsis

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive terbinafine hydrochloride cream applied on an ear pack. There is no comparator arm in this study.
Masking Description: Open-label design; neither participants nor investigators are blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Terbinafine Hydrochloride Cream (Experimental): Participants diagnosed with otomycosis will receive topical terbinafine hydrochloride cream applied on an ear pack. The pack will be inserted into the external auditory canal and changed every 2 days for a total duration of 2 weeks.
  Interventions: Drug: Terbinafine Hydrochloride Cream

INTERVENTIONS:
Drug: Terbinafine Hydrochloride Cream — Topical antifungal treatment. Terbinafine hydrochloride 1% cream will be applied on an ear pack, inserted into the external auditory canal, and changed every 2 days. Treatment continues for 14 days.

SUMMARY:
Otomycosis is a fungal infection of the ear that often causes itching, pain, ear discharge, and hearing problems. It is more common in hot and humid climates and in people with risk factors such as diabetes, frequent use of antibiotic ear drops, or swimming in polluted water. Standard treatments include antifungal ear drops, but relapses are frequent.

This study will evaluate the effectiveness of terbinafine hydrochloride cream, an antifungal medication, in treating otomycosis. Terbinafine is known to be active against fungi such as Aspergillus and Candida, which are common causes of ear fungal infections. In this study, patients with otomycosis will have terbinafine hydrochloride cream applied on an ear pack that will be placed in the ear canal and changed every two days for two weeks.

The main goal of the study is to find out whether terbinafine hydrochloride is effective in reducing symptoms and eradicating the fungal infection. Patients will be examined clinically and ear swabs will be tested before and after treatment. The study will be conducted at Assiut University Hospital and Assiut General Hospital in Egypt, and about 50 patients are expected to participate.

DETAILED DESCRIPTION:
Otomycosis is a common fungal infection of the external auditory canal. It is often associated with itching, ear blockage, tinnitus, pain, and hearing loss. Diagnosis is made clinically and confirmed by the presence of fungal growth on culture. Aspergillus species are the most frequent pathogens, but Candida species are also common.

Terbinafine hydrochloride is an antifungal drug from the allylamine class. It acts by inhibiting squalene epoxidase, an enzyme necessary for fungal cell membrane synthesis. Although terbinafine is not the first-line treatment for otomycosis, laboratory studies have shown it to be effective against Aspergillus and Candida, suggesting a potential role in therapy.

This single-arm, interventional clinical trial will include 50 patients diagnosed with otomycosis. Eligible participants will undergo full history and otoscopic examination. Ear swabs will be obtained before and after treatment for fungal culture. The intervention consists of applying terbinafine hydrochloride cream on an ear pack, which will be inserted into the ear canal. Packs will be replaced every two days for two weeks. Clinical follow-up will be performed at two weeks, and improvement will be assessed both by symptom relief and microbiological eradication.

The primary outcome is the percentage of patients who improve after terbinafine treatment. Secondary outcomes include symptom reduction and treatment safety. Data will be collected and analyzed using SPSS software. This study is approved by the Ethics Committee of the Faculty of Medicine, Assiut University. All patients will provide written informed consent prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (male or female).

Clinical diagnosis of otomycosis (presence of itching, ear discharge, ear canal debris, or fungal mass on otoscopic exam).

Confirmation of fungal infection by direct microscopy (KOH preparation) and/or culture.

Willingness to comply with study procedures and follow-up visits.

Provided written informed consent.

Exclusion Criteria:

* Age < 18 years.

Bacterial otitis externa, mixed bacterial-fungal infection, or chronic suppurative otitis media.

History of ear surgery or tympanic membrane perforation.

Use of systemic or topical antifungal agents within the last 2 weeks.

Known hypersensitivity or allergy to terbinafine or excipients of the study drug.

Immunocompromised patients (e.g., HIV/AIDS, chemotherapy, uncontrolled diabetes mellitus).

Pregnant or breastfeeding women.

Patients unable or unwilling to provide informed consent or adhere to treatment protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and mycological cure rate of otomycosis after topical terbinafine | 14 days (±3) from treatment initiation
  Proportion of participants achieving both: (a) clinical resolution of otomycosis signs and symptoms (itching, otalgia, otorrhea, canal edema/debris) with a normal otoscopic exam, and (b) negative fungal culture from an ear swab. "Cure" is defined as meeting both criteria; otherwise recorded as "no cure."
Clinical and mycological cure rate of otomycosis after topical terbinafine | 14 days (±3) from treatment initiation
  Proportion of participants achieving both: (a) clinical resolution of otomycosis signs and symptoms (itching, otalgia, otorrhea, canal edema/debris) with a normal otoscopic exam, and (b) negative fungal culture from an ear swab. "Cure" is defined as meeting both criteria; otherwise recorded as "no cure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478
- [Background] Hentzer E. Histologic studies of the normal mucosa in the middle ear, mastoid cavities and Eustachian tube. Ann Otol Rhinol Laryngol. 1970 Aug;79(4):825-33. doi: 10.1177/000348947007900414. No abstract available. PMID 5526992